CLINICAL TRIAL: NCT00816946
Title: Scaling up Evidence-based Nutrition Interventions to Address Maternal and Child Health Outcomes in Pakistan: a District-based Demonstration Project in Rural Sindh
Brief Title: District-based Mainstreaming Nutrition Project in Rural Pakistan
Acronym: NF Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); National Lady Health Workers Programme, Government of Pakistan (Unknown)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Director, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 753-Ped/ERC-07
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Malnutrition
Keywords: malnutrition; growth
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine LHW Advice (No Intervention): Arm receiving routine advice by their local Lady Health Workers (LHWs)
- Enhanced LHW Advice (Active Comparator): Arm receiving enhanced nutrition and health advice from the local Lady Health Workers (LHWs)during their routine community visits.
  Interventions: Behavioral: Enhanced education

INTERVENTIONS:
Behavioral: Enhanced education — Enhanced Nutritional education/counseling to mothers on the following topics:
  During Pregnancy: diet during pregnancy; antenatal care; iron tablets; colostrum Postpartum period: difficulties during lactation; diet during lactation; EBF; childhood vaccination; newborn care Complementary Feeding General Health: vitamin A; diarrhea management; iodine; hygiene for health; protection from malaria; ARI & protection against ARI
  Arms: Enhanced LHW Advice

SUMMARY:
This study aims to provide evidence regarding the feasibility of integrating an enhanced maternal and child care health education package into the existing curricula of the National Program for Family Planning and Primary Health Care (LHW Program) and evaluating the feasibility of scaling-up as well as the impact on birth outcomes, nutritional status, morbidity patterns and overall survival patterns at the community level.

DETAILED DESCRIPTION:
This project aims to do the following:

* To evaluate the operational feasibility of integrating an enhanced health education and nutrition package into the existing curriculum of the National Program for FP/PHC (LHW Program)
* Impact of the implementation of the full package of evidence-based nutrition interventions on the nutrition status, morbidity patterns and overall survival patterns in the district

ELIGIBILITY:
Inclusion Criteria:

* Live born infants and young children from all registered pregnancies within participating villages and catchment population
* pregnant women
* Consent given by at least one of the parents

Exclusion Criteria:

* Children born with congenital malformations or serious birth injury
* Suspected non-compliance (mobile and poorly motivated parents).
* Failure to give consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
mother pregnancy weight gain in 3rd trimester | at time of enrollment, 2 weeks before delivery
mothers Hb level | at time of enrollment, 2 weeks before delivery
child's birthweight | at birth

SECONDARY OUTCOMES:
young child's growth | 0, 3, 6, 12, 18 mths, at end of study
dietary diversity of CF | 6 mths, 9mths, 12mths, 18 mths

CONTACTS AND LOCATIONS:
Locations (1):
- AKU-Peds Naushero Feroze Site Office, Naushero Feroze, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No